CLINICAL TRIAL: NCT01969292
Title: Colometer - A Real Time Quality Improvement Feedback System for Screening Colonoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stage 1 Complete; Stage 2 and 3 not pursued
Sponsor: Christopher Andrews (Other)
Responsible Party: Sponsor-Investigator, Christopher Andrews, Associate Professor, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Col001
Record Dates: First submitted 2013-09-26; First posted 2013-10-25 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-01

CONDITIONS: Colon Cancer
Keywords: colonoscopy; quality assurance
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Colometer (Experimental): Colometer software will be engaged during the colonoscopy to provide real time feedback to the endoscopist.
  Interventions: Other: Colometer
- Sham Software (Sham Comparator): An identical set-up to the experimental arm but with a green band showing across the top for the duration of the colonoscopy.
  Interventions: Other: Sham Software
- Control (No Intervention): Recordings of colonoscopies made without Colometer or sham feedback during the course of the colonoscopy will be evaluated retrospectively using the Colometer software.

INTERVENTIONS:
Other: Colometer — Real time software based image analysis tool.
  Arms: Colometer
Other: Sham Software — Software that displays constant positive feedback that is unrelated to the quality measures of the actual colonoscopy.
  Arms: Sham Software

SUMMARY:
Our team has created an automated, real-time software based image analysis tool called Colometer to improve screening colonoscopy providing real time visual feedback on image quality. There are three components to this study. The first is to validate the bowel assessment preparation using the recorded colonoscopy videos from 50 consented normal risk patients. In the second phase, technological and machine user interface refinements will be identified and completed. Finally, the third phase will be a sham controlled prospective study of Colometer versus standard care in 100 consented average risk patients undergoing screening colonoscopy as performed by 10 consented endoscopists.

ELIGIBILITY:
Inclusion Criteria:

* Patients: patients categorized as normal risk who have been referred for screening colonoscopy at the Forzani & MacPhail Colon Cancer Screening Centre in Calgary, Alberta
* Endoscopists: Gastroenterologists with practices at the Forzani & MacPhail Colon Cancer Screening Centre, Calgary, Alberta

Exclusion Criteria:

* Patients: patients who are not categorized as normal risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
%Clear | Measurement will occur during the withdrawal phase as indicated by the physician during the colonoscopy procedure; on average, 12 minutes
  This is defined as the Percentage of the total withdrawal time where the withdrawal velocity is below a set speed limit and the view is clear (ie, not blurry) as measured by the software. Visualization of the colon lumen is ideal with a slow, non-blurry view in order to detect polyps.

SECONDARY OUTCOMES:
Average withdrawal velocity | Measurement will occur during the withdrawal phase as indicated by the physician during the colonoscopy procedure; on average, 12 minutes.
Ottawa Stool Score | Measurement will occur during the withdrawal phase as indicated by the physician during the colonoscopy procedure; on average, 12 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N Andrews, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- Forzani&MacPhail Colon Cancer Screening Centre, Calgary, Alberta, Canada